CLINICAL TRIAL: NCT06544304
Title: Interventional, Multicenter, Single-Arm Clinical Trial of Buttock Augmentation With Polymethylmethacrylate
Brief Title: Buttock Augmentation With Polymethylmethacrylate
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MTC MEDICAL COMERCIO INDUSTRIA IMPORTACAO E EXPORTACAO DE PRODUTOS BIOMEDICOS LTDA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MTC_01_2024_V1
Record Dates: First submitted 2024-07-31; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Aesthetics; Augmentation
Keywords: augmentation; gluteal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): PMMA (polymethylmethacrylate) 30% Biosimetric
  Interventions: Device: PMMA

INTERVENTIONS:
Device: PMMA — PMMA 30%

SUMMARY:
Single-arm multicenter interventional clinical trial of buttock augmentation with polymethyl methacrylate.

The objective is to evaluate the safety and effectiveness of using 30% Biosimetric PMMA gel for buttock augmentation.

DETAILED DESCRIPTION:
The sample will be 133 patients. Specific patients will be screened at study sites according to eligibility classifications. After signing the consent form, patients will be included in the study and will be monitored for 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years old;
* Signed Informed Consent Form (ICF);
* Participant understands and is willing to participate in the clinical study and attend visits.

Exclusion Criteria:

* Known history of allergy to formula components;
* Have the following morbidities (or any other disease that may interfere with the study): chronic inflammatory disease, immunosuppression, diabetes, hypertension, autoimmune disease, dermatological disease in the region to be treated, acute or chronic renal failure, history of coronary disease, history of cerebrovascular disease, current neoplasia, mental illness undergoing psychiatric treatment, obesity with a BMI above 30, asthma, bronchitis, seizures, hepatitis or other active infectious diseases;
* Pregnancy;
* Prior filling of glutes;
* Use of acetylsalicylic acid, anti-inflammatories, anticoagulants, in the fifteen days before the procedure.
* Vitamin D supplementation, with normal serum levels and which you do not agree to suspend;
* Use of anabolic hormones;
* Vitamin D (25 hydroxyvitamin D) greater than 70 ng/mL;
* Serum calcium greater than 10 mg/dL;
* Patients with total body PMMA volume of 650mL or more.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 133 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by clinical evaluation | Before application of PMMA and 6 and 9 months after the procedure
  Occurrence of adverse events in patients who underwent gluteal augmentation with 30% Biosymmetric PMMA. Expected events will be classified as adverse events when they persist for more than two weeks, and should be reported throughout the study. Adverse events not previously identified will also be monitored at all visits.

SECONDARY OUTCOMES:
Changes in normal values of laboratory biochemical tests | Before application of PMMA and 6 and 9 months after the procedure
  laboratory biochemical exams
Volumetric capacity of filled muscle assessed by ultrasound imaging | Before application of PMMA and 6 and 9 months after the procedure
  Using an ultrasound device, images of the gluteus will be obtained to analyze the thickness of the muscle, and thus estimate its volumetric capacity.
Physician satisfaction assessed by GAIS scale | Before application of PMMA and 4, 6 and 9 months after the procedure
  Physician satisfaction will be assessed using the Portuguese version of the Global Aesthetic Improvement Scale, assigning values according to the following parameters:
  Much improved (5): excellent cosmetic result after the procedure. Much improved (4): marked improvement in appearance from the initial condition, but not completely optimal for the patient.
  Better (3): obvious improvement in appearance from the initial condition. Unchanged (2): appearance is essentially the same as the original condition. Worse (1): appearance is worse than the original condition.
Patient satisfaction assessed by GAIS scale | Up to 4, 6 and 9 months after the procedure
  Patient satisfaction will be assessed using the Portuguese version of the Global Aesthetic Improvement Scale, assigning values according to the following parameters:
  Much improved (5): excellent cosmetic result after the procedure. Much improved (4): marked improvement in appearance from the initial condition, but not completely optimal for the patient.
  Better (3): obvious improvement in appearance from the initial condition. Unchanged (2): appearance is essentially the same as the original condition. Worse (1): appearance is worse than the original condition.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nicareta B, Pereira LH, Sterodimas A, Illouz YG. Autologous gluteal lipograft. Aesthetic Plast Surg. 2011 Apr;35(2):216-24. doi: 10.1007/s00266-010-9590-y. Epub 2010 Sep 25. PMID 20871994
- [Background] Talbot SG, Parrett BM, Yaremchuk MJ. Sepsis after autologous fat grafting. Plast Reconstr Surg. 2010 Oct;126(4):162e-164e. doi: 10.1097/PRS.0b013e3181ea4541. PMID 20885205
- [Background] Stojicic M, Jurisic M, Marinkovic M, Jovanovic M, Igic A, Nikolic Zivanovic M. Necrotizing Skin and Soft Tissue Infection after Gluteal Augmentation in a Perioperatively Asymptomatic COVID-19 Patient-Complications of the Post-Lockdown Era? A Case Report. Medicina (Kaunas). 2023 May 10;59(5):914. doi: 10.3390/medicina59050914. PMID 37241146
- [Background] Guzey S, Ergan Sahin A. Brazilian Butt Lift: An Experience Over 3000 Patients. Aesthetic Plast Surg. 2024 Jul;48(14):2677-2693. doi: 10.1007/s00266-024-03965-8. Epub 2024 Apr 5. PMID 38580866